CLINICAL TRIAL: NCT00295594
Title: An Open, Randomised, Multicenter, Clinical Study to Compare the Safety and Efficacy of Tacrolimus and Minimal Steroids in Combination With Either a Monoclonal Anti-IL2R Antibody (Daclizumab) or Mycophenolate Mofetil in Liver Allograft Transplantation.
Brief Title: Comparing Efficacy & Safety of Tacrolimus With/Without MMF or Monoclonal Anti-IL2R Antibody in Liver Transplantation.
Acronym: MARSILEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FG-506-01-27
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Liver Transplantation
Keywords: Tacrolimus; Liver Transplantation; Treatment Outcome; Immunosuppression
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: tacrolimus
- 2 (Experimental)
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — Immunosuppression
  Other Names: Prograf, FK506

SUMMARY:
To compare the efficacy and safety of two regimens containing tacrolimus and minimal steroids together with either monoclonal anti-IL2R antibodies (daclizumab) or mycophenolate mofetil.

DETAILED DESCRIPTION:
This prospective randomised trial which combines MMF with tacrolimus and so avoids steroids in immunosuppressive maintenance could demonstrate alternatives to current immunosuppressive regimens. There is evidence that reduced steroid usage could further decrease the onset of diabetes mellitus, hypertension and viral infections combined with high efficacy for patients and graft survival. Since the use of MMF in liver transplantation is becoming an alternative in the rescue setting this could contribute to a steroid-free immunosuppressive approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older who will undergo primary orthotopic liver or split liver allograft transplantation are eligible for the study. Patients receiving a liver transplant from cadaveric heart-beating donor with compatible AB0 blood type can be included.

Exclusion Criteria:

* Recipient of an auxiliary graft
* Patient is requiring initial sequential or parallel therapy with other immunosuppressive antibody preparation(s).
* Patient is requiring ongoing dosing with corticosteroids.
* Patient is exhibiting symptoms of, or is having any previous history of neoplastic disease
* Patient or donor is known to be HIV positive.
* Patient is allergic or intolerant to study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2005-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Incidence of and time to first biopsy proven acute rejection which requires treatment within 3 months following transplantation | 3 months

SECONDARY OUTCOMES:
Acute rejection. Incidence of and time to first acute rejection. Incidence of and time to first corticosteroid-resistant acute rejection. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Physician, Study Director — Astellas Pharma Europe B.V.
Locations (38):
- Belgium (3):
  - Ghent
  - Leuven
  - Liège
- Copenhagen, Denmark
- Helsinki, Finland
- Germany (7):
  - Bonn
  - Erlangen
  - Essen
  - Hamburg
  - Hanover
  - Kiel
  - Mainz
- Budapest, Hungary
- Italy (7):
  - Bari
  - Bergamo
  - Milan
  - Napoli
  - Padua
  - Palermo
  - Udine
- Poland (2):
  - Szczecin
  - Wroclaw
- Spain (10):
  - A Coruña
  - Barcelona
  - Córdoba
  - Granada
  - Madrid
  - Murcia
  - Pamplona
  - Santiago
  - Seville
  - Valencia
- Sweden (2):
  - Gothenburg
  - Uppsala
- Switzerland (2):
  - Bern
  - Zurich
- United Kingdom (2):
  - Leeds
  - Newcastle

REFERENCES:
- See also: Link to FDA website — http://www.accessdata.fda.gov/scripts/cder/drugsatfda